CLINICAL TRIAL: NCT05867550
Title: To Compare the Efficacy of (Rifaximin + Mebeverine), (Rifaximin + Amitriptyline), and (Rifaximin + Psyllium Husk) in Irritable Bowel Syndrome Associated With Diarrhea
Brief Title: To Compare the Efficacy of Drugs in Combination for Treating Irritable Bowel Syndrome Associated With Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Rashid Ali Khosa, Lecturer, Bahria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC 106/2022
Record Dates: First submitted 2023-04-04; First posted 2023-05-22 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome; Diarrhea; IBS-D
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — Rifaximin; mebeverine; Psyllium; Amitriptyline

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial in which participants will be divided into 3 treatment groups i.e. Group A, Group B and Group C.
  * Participants of Group A will receive drug combination of Rifaximin and Mebeverine
  * Participants of Group B will receive drug combination of Rifaximin and Amitriptyline
  * Participants of Group C will receive drug combination of Rifaximin and Psyllium Husk
  * Each group will be given a combination of drugs for 2 weeks
  Stool Frequency, Characteristic of Stool and Abdominal Pain will be assessed at day 0 and day 14 of intervention
  At the end of study period , efficacy of different drug combinations and their potential side effects will be compared between the treatment groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A ( Rifaximin + Mebeverine ) (Active Comparator): Tab. Rifaximin 550mg thrice daily per orally for 2 weeks
  Tab. Mebeverine 135mg twice daily per orally for 2 weeks
  Interventions: Drug: Rifaximin 550 MG; Drug: Mebeverine 135 MG
- Group B ( Rifaximin + Amitriptyline ) (Active Comparator): Tab. Rifaximin 550mg thrice daily per orally for 2 weeks
  Tab. Amitriptyline 25mg once daily per orally for 2 weeks
  Interventions: Drug: Rifaximin 550 MG; Drug: Amitriptyline Hydrochloride 25 MG
- Group C ( Rifaximin + Psyllium Husk ) (Active Comparator): Tab. Rifaximin 550mg thrice daily per orally for 2 weeks
  Psyllium Husk 15-30mg once daily per orally for 2 weeks
  Interventions: Drug: Rifaximin 550 MG; Drug: Psyllium Husk

INTERVENTIONS:
Drug: Rifaximin 550 MG — Rifaximin 550 MG Oral Thrice Daily for 2 weeks will be included in all three treatment regimes i.e A, B and C
  Other Names: Rifaxa 550MG; Nimixa 550 MG; Xifaxa 550MG; Zerifax 550MG; Nixaf 550 MG
Drug: Mebeverine 135 MG — Mebeverine 135 MG Oral Twice Daily for 2 weeks will be included in Group A Treatment Regimes
  Other Names: Colofac 135 MG; Spasler Neo 135 MG; Mebever 135 MG
  Arms: Group A ( Rifaximin + Mebeverine )
Drug: Psyllium Husk — Psyllium Husk 15-35 MG Oral Once Daily for 2 weeks will be included in Group C Treatment Regimes
  Other Names: Ispaghol
  Arms: Group C ( Rifaximin + Psyllium Husk )
Drug: Amitriptyline Hydrochloride 25 MG — Amitriptyline Hydrochloride 25 MG Oral Once Daily for 2 weeks will be included in Group B Treatment Regimes
  Other Names: Tryptanol 25 MG
  Arms: Group B ( Rifaximin + Amitriptyline )

SUMMARY:
The goal of this clinical trial is to compare the efficacy of four different drugs in combination for management of irritable bowel syndrome (IBS)-associated diarrhea. The main question to answer is:

* Is there a significant difference in effect of different drug combinations in management of irritable bowel syndrome with diarrhea?

Participants will be divided into 3 treatment groups.

* Each group will be given a combination of drugs for 2 weeks
* At the end of study, efficacy of different drug combinations and their potential side effects will be compared between the treatment groups

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare the efficacy of four different drugs (Rifaximin , Mebeverine, Amitriptyline and Psyllium Husk) in combination for management of irritable bowel syndrome (IBS)-associated diarrhea. The main question to answer is:

• Is there a significant difference in effect of different drug combinations in management of irritable bowel syndrome with diarrhea?

Total of 162 Participants will be enrolled in study.

* Participants will be divided into 3 treatment groups i.e. Group A, Group B and Group C.
* Participants of Group A will receive drug combination of Rifaximin and Mebeverine
* Participants of Group B will receive drug combination of Rifaximin and Amitriptyline
* Participants of Group C will receive drug combination of Rifaximin and Psyllium Husk
* Each group will be given a combination of drugs for 2 weeks

Stool Frequency, Characteristic of Stool and Abdominal Pain will be assessed at day 0 and day 14 of intervention

Data will be collected using Questionnaire. Questionnaire will be filled by the researcher

SPSS will be used for analysis of data and appropriate test like Chi square Test, Student T test and One way ANOVA will be used to draw conclusions about the efficacy of different drug combinations and their potential side effects between the treatment groups

ELIGIBILITY:
Inclusion Criteria:

Individual of both gender between the age of 18-50 years Diagnosed case of Irritable Bowel Syndrome associated with Diarrhea

Exclusion Criteria:

* Presence of co morbid diseases
* Coronary Artery Disease (CAD)
* Chronic Obstructive Pulmonary Disease (COPD)
* Congestive Heart Failure (CHF)
* Patients taking drugs which modify or aggravate symptoms of IBS (antidepressants, calcium channel blockers etc.)
* Patients having hyperthyroidism & gluten hypersensitivity
* Patients with alarming symptoms, viz. history of fever, passage of blood in stool, loss of weight, any organic gastrointestinal disease in the recent past
* Patients with recent change in bowel habits, patients on any other concomitant medication for abdominal pain, bowel disturbance or altering gastrointestinal motility and malignancy of any other organ
* Patients with Irritable Bowel Disease and Celiac disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Overall Improvement in Frequency of Diarrhea | 2 Weeks
  The study will assess change in number of stools per day from day 0 to day 14
Overall Improvement in Characteristic of Diarrhea | 2 Weeks
  The study will assess change in characteristic of stool type from type 6,7 to 4 according to Bristol Stool Chart from day 0 to day 14
Overall Improvement in Abdominal Pain | 2 Weeks
  The study will assess change in abdominal pain from day 0 to day 14
Compare Efficacy of Treatment Regimes in Treatment Groups | 4 Weeks
  The study will assess and compare the effect of each treatment regime on reduction of diarrhea, improvement in abdominal pain among the treatment groups

SECONDARY OUTCOMES:
To observe adverse effects of treatment regimes | 2 Weeks
  The study will observe number of participants with adverse effects like Nausea, Stomachache, Dizziness, Tiredness, Joint Pain, Headache, Heartburn, Constipation, Dry Mouth, Sedation and Bloating of drugs in different groups and compare them

CONTACTS AND LOCATIONS:
Overall Officials: Rashid Ali, Principal Investigator — Bahria University Health Science Campus Karachi
Locations (1):
- Bahria University Health Sciences Campus, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD data will be available 01 year after publication and will be available perpetually
Access Criteria: All the data will be assessable to all

REFERENCES:
- [Background] Alaqeel MK, Alowaimer NA, Alonezan AF, Almegbel NY, Alaujan FY. Prevalence of Irritable Bowel Syndrome and its Association with Anxiety among Medical Students at King Saud bin Abdulaziz University for Health Sciences in Riyadh. Pak J Med Sci. 2017 Jan-Feb;33(1):33-36. doi: 10.12669/pjms.331.12572. PMID 28367168
- [Background] Altomare A, Di Rosa C, Imperia E, Emerenziani S, Cicala M, Guarino MPL. Diarrhea Predominant-Irritable Bowel Syndrome (IBS-D): Effects of Different Nutritional Patterns on Intestinal Dysbiosis and Symptoms. Nutrients. 2021 Apr 29;13(5):1506. doi: 10.3390/nu13051506. PMID 33946961
- [Background] Axelrod CH, Saps M. The Role of Fiber in the Treatment of Functional Gastrointestinal Disorders in Children. Nutrients. 2018 Nov 3;10(11):1650. doi: 10.3390/nu10111650. PMID 30400292
- [Background] Bachani P, Kumar L, Kumar N, Fatima M, Naz S, Memon MK, Memon S, Rizwan A. Prevalence of Irritable Bowel Syndrome and Frequency of Symptoms in the General Population of Pakistan. Cureus. 2021 Jan 6;13(1):e12541. doi: 10.7759/cureus.12541. PMID 33564537
- [Background] Bai T, Xia J, Jiang Y, Cao H, Zhao Y, Zhang L, Wang H, Song J, Hou X. Comparison of the Rome IV and Rome III criteria for IBS diagnosis: A cross-sectional survey. J Gastroenterol Hepatol. 2017 May;32(5):1018-1025. doi: 10.1111/jgh.13642. PMID 27862281
- [Background] Barbara G, Cremon C, Azpiroz F. Probiotics in irritable bowel syndrome: Where are we? Neurogastroenterol Motil. 2018 Dec;30(12):e13513. doi: 10.1111/nmo.13513. PMID 30460770